CLINICAL TRIAL: NCT02166801
Title: A Small-step Program for Development of New Treatment Principles for Children With Cerebral Palsy and Other Neurodevelopmental Disorders
Brief Title: Small Step Intervention for Infants With Cerebral Palsy and Other Neurodevelopmental Disorders
Acronym: smallstep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Ann-Christin Eliasson, Professor, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Smallstep
Record Dates: First submitted 2014-06-12; First posted 2014-06-18 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Gross Motor Development Delay; Cerebral Palsy
Keywords: Cerebral palsy; Children; Early Intervention; Communication; Gross motor function; Hand function
MeSH Terms: conditions — Cerebral Palsy; Communication | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early intervention for infants (Active Comparator): A 30w intensive intervention according to the small step program, with daily practice sections conducted by parents at home, with weekly support by therapists.
  Interventions: Behavioral: Early intervention for infants
- Usual care (Active Comparator): Usual care means that the Children in this arm of the study participate in the established follow up program that is established at the Astrid Lindgrens Children's Hospital and offered to all Children that displays a delayed early gross and fine motor development.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: Early intervention for infants — Three foci are included in the intervention: Communication, Hand function and Mobility/gross motor function. The Hand & Cognition and Mobility steps will be conducted during two time-periods. Communication will have a separate one-time intervention at the start of the study (prior to step I) in addition to one intervention period during step III (figure 1). General principles for the small step program: Training will be conducted in the children's home by the parents on a daily basis. The families will get instructions and supervision in their home every week by the therapist responsible for each specific step of the intervention. For each focus there will be different steps using an adaptive logarithm for training, i.e., adapted to the functional level of the child aiming at the next small developmental step. The family will be actively involved in identifying new foci for practice.
  Arms: Early intervention for infants
Behavioral: usual care — Children displaying delayed development and at risk of developing cerebral palsy are continuously followed-up at the children's hospital. There are no strict rules for the frequency of appointments within the usual care program but the families typically meet a physiotherapist every third week during the first 2-3 months, thereafter about once a month. The frequency depends on the family's needs and wishes. If there is a continuous need for therapeutic intervention and need of contact with different professions, the families will be referred to the Habilitation Services when the child is between 8-12 months. The control group will follow this customary procedure in the hospital. The only difference will be the assessment procedure, the sessions with the speech pathologist and that they will get feedback of the children's progress after each examination.
  Arms: Usual care

SUMMARY:
Children with cerebral palsy (CP) have life-long motor disorders and are typically subjected to extensive treatment throughout childhood. Despite this there is a lack of evidence supporting the effectiveness of treatment aiming at improving motor function and activity in daily life. The primary area of interest of this research programme is to determine the effectiveness of an early intervention program in children younger than 12 months of age who are at risk of developing CP. A randomised control trial is planned, addressing hand use, mobility and communication in a home-based program. New treatment principles based on recent knowledge of brain plasticity will be employed.

The overarching goal of this research programme is to develop and evaluate new intervention principles for children with neurodevelopmental disorders based upon theories of early learning induced brain plasticity. Our overall aims can be formulated as follows:

To evaluate the effects of an early intervention programme on the overall development in children with risk of developing cerebral palsy and other neurodevelopmental disorders. The program includes intensive intervention towards the foci: hand use, mobility and communication in a home based program

The hypothesis is that the design of the Small-Step-Program intervention, with clear foci on specific areas of development during different time periods and conducted in the child's home environment, will facilitate development and be more effective than usual care.

The second hypothesis is that children learn what they practice, meaning that children will have a more rapid development within the focus of each specific step in the training, when compared to the, for the time being, untrained steps.

The third hypothesis is that children's ability to learn within the different steps of the intervention programme will be influenced by the specific characteristics of any underlying brain pathology.

The fourth hypothesis is that parents in the study group will be less stressed and can better cope with their child's situation than parents to children receiving usual care. Thus, the tools provided within the Small-Step-Program intervention, like education, supervision and feedback of how to practice communication and task performance will make parents more able to cope with the child's delayed development.

DETAILED DESCRIPTION:
Rational for subject selection: Signs of CP may be visible already during the first months, but according to recommendations the diagnosis of CP should typically not be made until 2-4 years of age. The reason is that the individual developmental trajectories of muscle tone, postural control and motor function vary considerably during the first two years. A child with a late development may recover and atypical signs may disappear, and opposite, CP may develop although there have been no early signs. Thus, there is a dilemma in that it is too late to wait with early intervention until the CP diagnosis has been made. In this project we are addressing this problem by developing criteria for infants with high risk to develop CP based on early signs of atypical motor development and on perinatal risk factors. That means that we will include both infants who will get and infants who will not get the CP diagnosis. Children who are not meeting the criteria of CP at 2 years of age will be excluded from the analysis. The investigators assume that the intervention will influence the course of development and help the children to function at a higher level, but not that the intervention will "cure" CP and prevent later diagnosis. Infants with increased risk to develop CP will be recruited in this project.

The study group will be recruited from infants exposed to increased perinatal risk factors, such as preterm birth, hypoxia, infections, retinopathy of prematurity (ROP) chronic lung disease and heart insufficiency, small for gestational age, hypoxic ischemic insult and morphological brain abnormalities. These children commonly participate in a clinical follow up programme at the children's hospital with regular examinations at 3months. The high-risk preterm infants that at follow up examinations exhibit a delayed psycho-motor development or display clinical signs of abnormal neurology will be recruited. Recruitment will also include children below 8 months, demonstrating delayed psycho-motor development or clinical signs of abnormal neurology referred to the physiotherapy department from child neurologists at the hospital.

Randomisation The aim is to include 40 children in the study group with neurodevelopmental disorder to reach sufficient power in the study. This number is high but the investigators expect that about 50% will not fulfil the diagnose criteria at 2 years of age based on previous experience from intervention studies. The aim is to include 20 children with CP, which is a reasonable approximation of study population size to reach sufficient power. The children will be allocated to group by block randomisation. The intervention group (n=20) will take part in a newly developed Small-Step-Program. The comparison group (n=20) will continue their ordinary follow up programme. Stratification will be used to control for gestational age (preterm<37 and term>37 week). Children in the Small-Step-Program" will be further randomised to start with the mobility step or hand use step.

Rational for second randomisation Our hypothesis is that the trained step will improve, while the non-trained step will result in minor changes and that children in the control group will have a continuous developmental pace. The randomised steps are hand use and mobility.

The children in both groups will be assessed at four occasions, at start (first examination), after 12 weeks (second examination) and after 30 weeks (third examination) as well as at 2 years of age (fourth examination). For children in the study group there will be 3 additional times for assessments in order to investigate the second hypothesis. Parents in both groups will be asked to fill in questionnaires' at all four examinations. Both parents will be asked to fill out the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

will be based on delayed psychomotor development, as assessed by Alberta Motor Infants Scale, using -2SD as a cut-off point. Neurological signs will be investigated by Hammersmith Infant Neurological examination (HINE) together with a clinical neurological examinations. Magnetic resonance imaging (MR) will be used if available to support the risk of development of CP, only MR done for clinical purpose will be used. The risk factors suggested for inclusion in the intervention program will be confirmed by a child neurologist.

Exclusion Criteria:

is unstable health, uncontrolled epilepsy, progressive disorder, diagnosis with a specific syndrome. Parent's communication language should be Swedish or English with satisfactory skills in either language for simple conversation. If the children show a catch-up in development at the second assessment (after 12 weeks) and show no sign of neurodevelopmental disorder the program will be terminated

Ages: 4 Months to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales (PDMS-2) is used to measure change over time | Small Step group: at baseline, 6w, 12w,18w, 24w, 30w and 2 years. In the usual care group: at baseline, 12 w, 30w and at 2 years.
  Assesses gross and fine motor skills in young children. It is designed to evaluate children from birth through age 5. The PDMS-2 is composed of six subtests that assess related motor abilities that develop early in life: Reflexes, Stationary (body control and equilibrium), Locomotion, Object Manipulation, Grasping, and Visual-Motor Integration. Results from these subtests are used to generate the three composite scores: Gross Motor Quotient, Fine Motor Quotient, and Total Motor Quotient. Scores are presented as percentiles, standard scores, and age equivalents. Norms, based on a nationally representative sample of more than 2,000 children, are stratified by age

SECONDARY OUTCOMES:
Alberta Infant Motor Scale (AIMS) is used to measure change over time | Small Step group: at baseline, 6w, 12w,18w, 24w, 30w and 2 years. In the usual care group: at baseline, 12 w, 30w and at 2 years.
  Identifies infants who are delayed or deviant in motor development. It can be used from birth through independent walking (0-18 months). It identifies the gross motor performance of an infant compared to norm- referenced sample. It is an observational assessment and is quick to administrate with limited handling. The focus is on milestones and quality of posture and movement.
Hand Assessment for Infants, (HAI) is used to measure change over time | Small Step group: at baseline, 6w, 12w,18w, 24w, 30w and 2 years. In the usual care group: at baseline, 12 w, 30w and at 2 years.
  HAI is developed to identify and measure upper limb asymmetry and general manual development from 3-12 month in children at risk of developing cerebral palsy. During the test procedure, the aim is to elicit goal-directed functional use of the hands by introducing toys to be explored with both a uni-manual and a bimanual approach.
Gross Motor Function Measure (GMFM-66) is used to measure change over time | Small Step group: at baseline, 6w, 12w,18w, 24w, 30w and 2 years. In the usual care group: at baseline, 12 w, 30w and at 2 years.
  Gross Motor Function Measure (GMFM-66), is an observational, standardized and criterion-referenced measure, developed to evaluate change in gross motor function in children with cerebral palsy. The items cover gross motor capacity from lying and rolling, to walking, running and jumping.
Hammersmith Infant Neurological Examination (HINE) is used to measure change over time | Small Step group: at baseline, 6w, 12w,18w, 24w, 30w and 2 years. In the usual care group: at baseline, 12 w, 30w and at 2 years.
  HINE is a method to estimate the neurological development of infants aged two-24 month. Using HINE, the risk of neural disorder can be assessed.
Bayley Scales of Infant Development (BSID-III) is used to measure change over time | Two occacions in both groups: 30w and 2 years.
  is a standard measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers, ages 0-3. This measure consists of a series of developmental play tasks and takes between 45 - 60 minutes to administer. Raw scores of successfully completed items are converted to scale scores and to composite scores. These scores are used to determine the child's performance compared with norms taken from typically developing children of their age (in months).
Responsive Augmentative and Alternative Communication Style Scale (RAACS) is used to measure change over time | Small Step group: at baseline, 12w,18w, 30w and 2 years. In the usual care group: at baseline, 12 w, 30w and at 2 years.
  RAACS was developed for the purpose of assessing parents' communicative styles with children with communication difficulties. It is a video film of free communication between parents and children of maximum of 10 minutes. It is a criterion based assessment in which the films should be coded on 7 domains on a three grading scale. The results from the Responsive Augmentative and Alternative Communication Style Scale (RAACS) Version 3 can be used for planning and intervention as well as an outcome measure.
Swedish Parenthood Stress Questionnaire (SPSQ) is used to measure change over time | Both groups: baseline, 12w, 30w and at 2 years
  SPSQ measures perceived parental stress and is a revised version of the parent domain of the Parenting Stress Index. The instrument contains 34 items within the five sub-areas: Incompetence regarding parenthood, Role restriction, Social isolation, Spouse relationship problems, and Health problems.
The Hospital Anxiety and Depression Scale (HADS) is used to measure change over time | Both groups: baseline, 12w, 30w and at 2 years
  HADS is a self-assessment scale, was developed to detect states of depression, anxiety and emotional distress amongst patients who were being treated for a variety of clinical problems. The Swedish version of the instrument will be used.
The Working Model of the Child Interview, (WMCI) is used to measure change over time | Both groups: 30w and 2 years
  The WMCI is semi-structured, open-ended interview designed to assess parent´s representations of their infant/ child and their relationship with their infant/ child. The interview is video-taped and takes approximately one hour. The WMCI is coded and summarized in classification types reflecting the parents´ overall state of mind with respect to the relationship with the infant /child. WMCI has been found to be both a reliable and valid approach to scoring representational aspects of parent-child-relationships.
Swedish Early Communicative Development Inventory, SECDI is used to measure change over time | Both groups: 30w and 2 years
  parent questionnaire. SECDI is the Swedish version of The MacArthur Communicative Development Inventories, CDI. CDI is an internationally recognized parent report instrument for assessing early language development of children. The reliability and validity of The Swedish version of CDI, Swedish Early Communication Development Inventory (SECDI) have been investigated thoroughly and have been found to be satisfying. The instrument consists of two separate inventories: Words and gestures (CDI/WG) for children eight to 16 months and Words and Sentences (CDI/WS) for children 16 to 30 months. The SECDI inventories involve questions about communication and language capacities corresponding to the child's ability to comprehend and use communication and language.
Parent-Child Early Relational Assessment, PC-ERA is used to measure change over time | Both groups: 30w and 2 years
  Parent-Child Early Relational Assessment, PC-ERA. The PC-ERA measures parent´s and child´s affect and behavioral characteristics using parent items, child items as well as dyadic items. Ratings are based on observations of videotaped parent-child interactions in three types of situations; free play, feeding and structured task. The purpose of the method is to capture the child´s experience of the parent, the parents 'experience of the child, the affective and behavioral characteristics that each bring into the interaction, and the quality or tone of the relationship. PC-ERA has been used internationally, and reliability and validity of the method have been addressed in both high-risk and normative populations with positive outcomes.
Pediatric Evaluation of the Disability Inventory (PEDI) is used to measure change over time | Both groups: 30w and 2 years
  is a norm and criterion-referenced measure which evaluates functional skills and caregiver assistance in the domains self-care, mobility, and social function(17). The child is assessed by structured interviews with the parents. The summary scores can be converted to normative standard scores and scaled scores. The normative score are available for children 6 month to 7.5 years. The scaled scores range on a continuum from 0 to 100, where 0 represents no ability and 100 represents full capability to perform the functional skill items in a particular domain. PEDI is available in a Swedish version.
Parent Development Interview, PDI-R is used to measure change over time | 2 occacions in both groups, after intervention and at 2 year follow up
  is a semi-structured clinical interview intended to examine parents' representations of their children, themselves as parents, and their relationships with their children. The reliability and validity of the method has been considered good

OTHER OUTCOMES:
Semi structured interview | After interventionprogram, 30w, in the Small step group
  Semi structured interview measuring the parent's views of the feasibility and effectiveness of the Small Step program
Structural magnetic resonance imaging (MRI) | One time when the child is approximately 10-24 months
  It is well established that the timing, extent and characteristics of the underlying brain lesion in the children that will develop CP influence long-term motor development. However, little is known about how specific lesion characteristics influence the outcome of early intervention. It is now common practice to include a structural MRI, including diffusion sequences, of the brain in the diagnosis process for children that are at risk of developing CP in Sweden. The information about the underlying lesion from this MRI examination is essential to investigate the fourth hypothesis of this study. A copy of the images from the clinical MRI will be collected at the time when the scan is performed. This means that the children included in the project will not undergo any extra structural MRI examinations outside the normal clinical routine. Neuroimaging data will be assessed by experienced neuroradiologists in accordance with well established clinical assessment protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Astrid Lindgren Children Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Eliasson AC, Holmstrom L, Aarne P, Nakeva von Mentzer C, Weiland AL, Sjostrand L, Forssberg H, Tedroff K, Lowing K. Efficacy of the small step program in a randomised controlled trial for infants below age 12 months with clinical signs of CP; a study protocol. BMC Pediatr. 2016 Nov 3;16(1):175. doi: 10.1186/s12887-016-0711-x. PMID 27809886